CLINICAL TRIAL: NCT01426802
Title: A 12 Week Multi Center, Open Label, Single Arm Study to Assess the Safety and Efficacy of Vildagliptin 50 mg Twice Daily in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin
Brief Title: Vildagliptin 50 mg Twice Daily in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AEG01
Record Dates: First submitted 2011-07-01; First posted 2011-08-31 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: metformin; vildagliptin; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

ARMS (1):
- Vildagliptin 50 bid (Experimental)
  Interventions: Drug: vildagliptin

INTERVENTIONS:
Drug: vildagliptin — Drug 50mg vildagliptin bid

SUMMARY:
The study is designed to demonstrate the short term efficacy and safety of vildagliptin 50 mg bid in patients with Type 2 Diabetes Mellitus inadequately controlled with Metformin.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the informed consent
* HbA1c in the range of > 7 to ≤10.5% at Visit 1
* Ability to comply with all study requirements

Exclusion Criteria:

* Pregnant or lactating women
* Serious cardiovascular disorders
* Liver/renal disease or dysfunction
* Anti-diabetic other than metformin, thiazolidine, or α-GI or insulin
* Laboratories values abnormalities as defined by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of vildagliptin 50 mg bid | 12 weeks
  Efficacy of vildagliptin based on the reduction in mean HbA1c and mean fasting plasma glucose with vildagliptin treatment at 12 weeks. Safety is measured by monitoring lipids profile, liver and kidney function to assess vildagliptin safety.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Investigative site, Cairo, Egypt